CLINICAL TRIAL: NCT06423027
Title: Exploring the Influence of Nature-Oriented Chatbots on the Mental Health of Older Adults Living Alone
Brief Title: Nature-Oriented Chatbots on Older Adults' Mental Health
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: N202403042
Record Dates: First submitted 2024-05-08; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-04

CONDITIONS: Depression; Loneliness; Happiness; Connection With Nature; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Experiment (Experimental)
  Interventions: Behavioral: Nature-Oriented Chatbots

INTERVENTIONS:
Behavioral: Nature-Oriented Chatbots — Nature-oriented chatbots are an intervention with nature-based video delivered by self-developed chatbots
  Arms: Experiment

SUMMARY:
This study aims to explore the influence of nature-oriented chatbots on the mental health of older adults residing alone. Leveraging the therapeutic potential of nature exposure and the interactive capabilities of chatbot technology, our research seeks to investigate whether engaging with nature-oriented chatbots can mitigate feelings of depression, and loneliness while enhancing overall psychological well-being and quality of life. Through a combination of experimental interventions and psychological assessments, the investigators will assess the impact of nature-oriented chatbots on participants' mental health outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 60 years and above who live alone.
2. Regular users of smartphones, with internet access, and proficient in using LINE.
3. Individuals who consent to participate in the study and sign the consent form.
4. Capable of understanding interactive messages and the content of pre- and post-test questionnaires.

Exclusion Criteria:

1. Individuals without smartphones, internet access, or not using LINE.
2. Diagnosed with sensory impairments.
3. Diagnosed with mental illnesses requiring continuous treatment.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Depression | up to 8 weeks
  The Geriatric Depression Scale
loneliness | up to 8 weeks
  UCLA loneliness (ULS-8)
happiness | up to 8 weeks
  Well-being of Older People measure (WOOP)
connection with nature | up to 8 weeks
  Connectedness with nature scale (CNS）